CLINICAL TRIAL: NCT03694548
Title: Acceptability, Feasibility and Safety of a Yoga Program for Chronic Pain in Sickle Cell Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to COVID-19 pandemic.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nitya Bakshi, Assistant Professor of Pediatrics, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00102878
Record Dates: First submitted 2018-09-25; First posted 2018-10-03 (Actual); Results first posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Sickle Cell Disease
Keywords: Yoga; Behavioral/Social; Pediatrics
MeSH Terms: conditions — Anemia, Sickle Cell; Behavior

STUDY DESIGN:
Intervention Model Description: Part A: Survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of yoga program in adolescent patients with SCD and chronic pain and their parents
  Part B: Feasibility and safety of yoga program in adolescent patients with SCD and chronic pain from Part A
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A Survey: Group 1 Adolescent Patients with SCD (Other): Adolescent patients with SCD and chronic pain completed a survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program for chronic pain in SCD.
  Interventions: Behavioral: Part A Survey
- Part A Survey: Group 2 Parents of Adolescent Patients with SCD in Part A (Other): Parents of adolescent patients with SCD and chronic pain from Group 1 completed a survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program for chronic pain in SCD.
  Interventions: Behavioral: Part A Survey
- Part B Yoga Program (Experimental): Participants from Part A Group 1 had the opportunity to enroll in Part B to receive eight in-person instructor-led group yoga sessions.
  Interventions: Behavioral: Part B Yoga Program

INTERVENTIONS:
Behavioral: Part A Survey — Survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program for chronic pain in SCD.
  Arms: Part A Survey: Group 1 Adolescent Patients with SCD; Part A Survey: Group 2 Parents of Adolescent Patients with SCD in Part A
Behavioral: Part B Yoga Program — Eight in-person instructor-led group yoga sessions.
  Arms: Part B Yoga Program

SUMMARY:
Chronic Pain is associated with morbidity and poor quality of life in patients with Sickle Cell Disease (SCD). Complementary therapies, such as yoga are beneficial in patients with non-SCD chronic pain conditions. Yoga was shown to be acceptable, feasible and helpful in one study in acute SCD pain. The purpose of the study is to assess the acceptability, feasibility, and safety of yoga for chronic pain in SCD.

DETAILED DESCRIPTION:
Pain is a major cause of morbidity, impaired quality of life, and healthcare utilization in SCD. Yoga is beneficial in patients with non-SCD chronic pain conditions. Yoga was shown to be acceptable, feasible and helpful in one study in acute SCD pain, but there are currently no data on yoga for chronic pain in SCD.

This study has the following aims:

In Aim 1, the study will assess the acceptability of yoga for chronic pain in SCD. The study will also assess the feasibility and safety of a yoga program for adolescents with SCD and chronic pain.

In Aim 2, the study will study the feasibility of collection of psychological and patient-reported outcomes in a study of yoga for chronic pain in SCD.

In Aim 3, the study will explore patient acceptability of yoga and conduct a needs assessment for the development of a smartphone app for yoga through qualitative interviews.

This study will be conducted in 2 parts, Part A and Part B:

Part A will assess attitudes and practices related to yoga and potential acceptability of a yoga program in adolescents with SCD and chronic pain (Group 1), and their parents/guardians (Group 2). Up to 40 adolescents who meet inclusion criteria, and do not meet exclusion criteria, and their parent/guardian will be enrolled on Part A until 20 adolescents are enrolled on Part B. Only one parent/guardian per adolescent participant will be enrolled.

Part B will assess the feasibility and safety of a yoga program for SCD and chronic pain. This program will comprise of 8 instructor-led group yoga sessions. The study will measure psychological factors implicated in chronic pain, and pain-related patient-reported outcomes, and assess the feasibility of collection of these outcomes. The study will also explore patient acceptability of yoga through qualitative interviews and conduct a needs assessment for the development of a smartphone app for yoga. Up to 20 adolescents who meet inclusion criteria, and do not meet exclusion criteria will be enrolled in Part B.

ELIGIBILITY:
Inclusion Criteria:

* SCD, any genotype
* Presence of chronic pain, the presence of chronic pain will be defined based on the frequency characteristic of the Analgesic, Anesthetic, and Addiction Clinical Trial Translations Innovations Opportunities and Networks (ACTTION)-American Pain Society Pain Taxonomy (AAPT) criteria for chronic SCD pain, as the presence of SCD-related pain on 15 or more days of the month, for the past 6 months
* Age 12 -21 at time of enrollment
* English speaking

Exclusion Criteria:

* Daytime or nighttime oxygen requirement for hypoxia
* Most recent hemoglobin < 5 or platelet count < 20
* Known pregnancy
* Severe cognitive issues not allowing for understanding consent/assent and instructions
* History of overt stroke with significant residual motor weakness
* History of recurrent syncope
* Any other comorbidities or health concerns that the treating healthcare provider or investigators feel are a contra-indication for participation in the study

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitya Bakshi, MBBS, MS, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bakshi N, Cooley A, Ross D, Hawkins L, Sullivan M, Astles R, Sinha C, Katoch D, Peddineni M, Gee BE, Lane PA, Krishnamurti L. A pilot study of the acceptability, feasibility and safety of yoga for chronic pain in sickle cell disease. Complement Ther Med. 2021 Jun;59:102722. doi: 10.1016/j.ctim.2021.102722. Epub 2021 Apr 21. PMID 33892094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the trial was between October 2018 and March 2020.
Pre-assignment Details: In Part A of this two-part study, adolescents with SCD and chronic pain (Group 1) and their parent (Group 2) completed a survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program for chronic pain in SCD. In Part B, the study assessed the feasibility and safety of an instructor-led group yoga program.
Groups:
- Part A Survey Adolescent Patients With SCD and Chronic Pain (Group 1): Adolescent patients with Sickle Cell Disease (SCD) and chronic pain completed a survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program for chronic pain in SCD.
  Part A Survey: Survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program for chronic pain in SCD.
- Part A Survey Parents of Patients in Part A (Group 2): Parents of adolescent patients with SCD and chronic pain from Group 1 completed a survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program for chronic pain in SCD.
  Part A Survey: Survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program for chronic pain in SCD.
- Part B Yoga Program: Participants from Part A Group 1 had the opportunity to enroll in Part B to receive eight in-person instructor-led group yoga sessions.
  Part B Yoga Sessions: Eight in-person instructor-led group yoga sessions.
Period: Part A Survey
Arm/Group | Part A Survey Adolescent Patients With SCD and Chronic Pain (Group 1) | Part A Survey Parents of Patients in Part A (Group 2) | Part B Yoga Program
Started | 18 | 17 | 0
Completed | 15 | 14 | 0
Not Completed | 3 | 3 | 0
Not completed — Protocol Violation | 3 | 3 | 0
Period: Part B Yoga Program
Arm/Group | Part A Survey Adolescent Patients With SCD and Chronic Pain (Group 1) | Part A Survey Parents of Patients in Part A (Group 2) | Part B Yoga Program
Started | 0 | 0 | 12
Completed | 0 | 0 | 1
Not Completed | 0 | 0 | 11
Not completed — Protocol Violation | 0 | 0 | 3
Not completed — Did not attend intervention | 0 | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Part A & B Adolescent Patients With SCD and Chronic Pain: Part A: Adolescent patients with sickle cell disease (SCD) and chronic pain completed a survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program.
  Part B: Part A adolescent patients with SCD then had the opportunity to enroll in Part B yoga program.
- Parents of Patients in Part A (Group 2): Parents of patients in Part A completed a survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program.
- Total: Total of all reporting groups
Arm/Group | Part A & B Adolescent Patients With SCD and Chronic Pain | Parents of Patients in Part A (Group 2) | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Parents were not enrolled in Part B. 12 participants started Part B, but only 9 participants are included as the number analyzed because 3 subjects were withdrawn due to protocol violation and not analyzable.
  years
    Part A | 16 [14 to 17] | 43.5 [42 to 51] | 18 [16 to 43]
    Part B: number analyzed (Participants) | 9 | 0 | 9
    Part B | 17 [15 to 18] |  | 17 [15 to 18]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Parents were not enrolled in Part B. 12 participants started Part B, but only 9 participants are included as the number analyzed because 3 subjects were withdrawn due to protocol violation and not analyzable.
  Participants
    Part A: Female | 8 | 13 | 21
    Part A: Male | 7 | 1 | 8
    Part B: number analyzed (Participants) | 9 | 0 | 9
    Part B: Female | 5 | 0 | 5
    Part B: Male | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Parents were not enrolled in Part B. 12 participants started Part B, but only 9 participants are included as the number analyzed because 3 subjects were withdrawn due to protocol violation and not analyzable.
  Participants
    Part A: American Indian or Alaska Native | 0 | 0 | 0
    Part A: Asian | 0 | 0 | 0
    Part A: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Part A: Black or African American | 12 | 12 | 24
    Part A: White | 0 | 1 | 1
    Part A: More than one race | 3 | 1 | 4
    Part A: Unknown or Not Reported | 0 | 0 | 0
    Part B: number analyzed (Participants) | 9 | 0 | 9
    Part B: American Indian or Alaska Native | 0 | 0 | 0
    Part B: Asian | 0 | 0 | 0
    Part B: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Part B: Black or African American | 7 | 0 | 7
    Part B: White | 0 | 0 | 0
    Part B: More than one race | 2 | 0 | 2
    Part B: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number (Proportion) of Adolescent Patients With SCD and Chronic Pain Approached That Consent to Participate in Part A
Description: The study hypothesis that the proportion of adolescent patients with SCD and chronic pain approached that consent to complete a survey to assess attitudes and practices related to yoga (Part A) will be 50% or greater.
Time Frame: Enrollment visit
Population: Unable to assess outcome: As eligibility for Part A was determined based on patient response regarding presence of chronic pain, and if patients were not interested when approached to determine eligibility or potential interest in the study, we were not always able to assess if they would have met eligibility criteria. Thus, we were not able to accurately estimate the proportion of individuals with SCD and chronic pain who agreed to participate in Part A.
Groups:
- Part A Survey Adolescent Patients With SCD and Chronic Pain: Adolescent Patients with Sickle Cell Disease (SCD) and chronic pain completed a survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program.
  Part A Survey: Survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program.
Arm/Group | Part A Survey Adolescent Patients With SCD and Chronic Pain
Number analyzed (Participants) | 0

2. Primary Outcome: Number (Proportion) of Adolescent Patients With SCD and Chronic Pain Enrolled in Part A That Consent to Participate in Part B
Description: The study hypothesis is that the proportion of adolescent patients with SCD and chronic pain enrolled in Part A that consent to participate in Part B will be 50% or greater.
Time Frame: Enrollment visit
Measure: Count of Participants; unit: Participants
Groups:
- Part A Survey Adolescent Patients With SCD and Chronic Pain: Part A: Adolescent Patients with Sickle Cell Disease (SCD) and chronic pain completed a survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program.
  Participants from Part A Group 1 had the opportunity to enroll in Part B to receive eight in-person instructor-led group yoga sessions. Part B Yoga Sessions: Eight in-person instructor-led group yoga sessions.
Arm/Group | Part A Survey Adolescent Patients With SCD and Chronic Pain
Number analyzed (Participants) | 18
Participants | 12

3. Primary Outcome: Number (Proportion) of Participants Enrolled in Part B That Attend at Least 6 of 8 Yoga Sessions.
Description: The study hypothesis is that the proportion of participants enrolled in Part B that attend at least 6 of 8 in-person yoga sessions will be 80% or greater.
Time Frame: Through study completion, up to one year
Population: 12 participants started Part B, but only 9 participants are included as the number analyzed because 3 subjects were withdrawn due to protocol violation and not analyzable.
Measure: Count of Participants; unit: Participants
Groups:
- Part B Yoga Program: Participants enrolled in Part B will receive eight in-person instructor-led group yoga sessions.
  Yoga program: Instructor-led group yoga sessions (Part B): Participants enrolled in Part B will receive eight in-person instructor-led group yoga sessions. Proposed yoga session will comprise of poses, breathing exercises, and guided relaxation.
Arm/Group | Part B Yoga Program
Number analyzed (Participants) | 9
Participants | 0

4. Primary Outcome: Number (Proportion) of Participants Enrolled in Part B With an Emergency Department Visit or a Hospitalization for Pain Within 24 Hours of Completion of Each Yoga Session.
Description: The study hypothesis is that the proportion of participants enrolled in Part B with an Emergency Department visit or a hospitalization for pain within 24 hours of completion of each yoga session will be 30% or less.
Time Frame: Through study completion, up to one year
Population: Only assessed in participants who were able to attend yoga sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Yoga Program
Number analyzed (Participants) | 1
Participants | 0

5. Primary Outcome: Number (Proportion) of Participants in Part B Who Complete All Study Assessments Before, and at the End of the Yoga Program.
Description: The study hypothesis is that the proportion of participants who complete all study assessments before, and at the end of the yoga program will be 70% or greater.
Time Frame: Through study completion, up to one year
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Yoga Program
Number analyzed (Participants) | 1
Participants | 0

6. Primary Outcome: Adherence to Submission of Pain Diary (Number/Proportion of Participants Who Submit at Least 4 Days of Pain Diary Data Before, and at the End of the Yoga Program)
Description: The study hypothesis is that the proportion of participants who submit at least 4 days of pain diary data before, and at the end of the yoga program will be 70% or greater.
Time Frame: Through study completion, up to one year
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Yoga Program
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: Through study completion, up to one year.
Groups:
- Part A Group 1: Adolescent SCD Patients Survey: Adolescent Sickle Cell Disease (SCD) Patients with chronic pain completed a survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program.
  Part A Survey: Survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program.
- Part A Group 2: Parents of Adolescent SCD Patients Survey: Parents of adolescent SCD Patients with chronic pain from Group 1 completed a survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program.
  Part A Survey: Survey designed to capture pain characteristics, attitudes and practices related to yoga, and potential acceptability of a yoga program.
- Part B Adolescent SCD Patients Yoga Program: Participants from Part A Group 1 had the opportunity to enroll in Part B to receive eight in-person instructor-led group yoga sessions. Part B Yoga Sessions: Eight in-person instructor-led group yoga sessions.
Arm/Group | Part A Group 1: Adolescent SCD Patients Survey | Part A Group 2: Parents of Adolescent SCD Patients Survey | Part B Adolescent SCD Patients Yoga Program
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/9
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/9

LIMITATIONS AND CAVEATS:
See published manuscript

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT03694548/Prot_SAP_000.pdf